CLINICAL TRIAL: NCT00162123
Title: A Multi-Center, Open-Label, Phase II Study of Ipilimumab (MDX-010 Extended-Treatment Monotherapy or Follow-up for Patients Previously Enrolled in Ipilimumab (MDX-010) Protocols.
Brief Title: A Companion Study for Patients Enrolled in Prior/Parent Ipilimumab Studies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-025
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: Melanoma
Keywords: ipilimumab; previously treated
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- First reinduction: Ipilimumab, 0.3 to 10 mg/kg (Experimental): Participants who initially received ipilimumab, 0.3 mg/kg, in a parent study received ipilimumab, 10 mg/kg in the current study. Ipilimumab was administered as an individual open-label dose every 3 weeks for the first 10 weeks of reinduction for a total of 4 separate doses unless the patient experienced disease progression or withdrew consent. Participants had to wait 3 weeks from the last dose of ipilimumab in a parent study to the first dose of ipilimumab in the current study.
  Interventions: Drug: Ipilimumab
- First reinduction: Ipilimumab, 3 to 10 mg/kg (Experimental): Participants who initially received ipilimumab, 3 mg/kg, in a parent study received ipilimumab, 10 mg/kg in the current study. Ipilimumab was administered as an individual open-label dose every 3 weeks for the first 10 weeks of reinduction for a total of 4 separate doses unless the patient experienced disease progression or withdrew consent. Participants had to wait 3 weeks from the last dose of ipilimumab in a parent study to the first dose of ipilimumab in the current study.
  Interventions: Drug: Ipilimumab
- First reinduction: Ipilimumab, 10 to 10 mg/kg (Experimental): Participants who initially received ipilimumab, 10 mg/kg, in a parent study received ipilimumab, 10 mg/kg in the current study. Ipilimumab was administered as an individual open-label dose every 3 weeks for the first 10 weeks of reinduction for a total of 4 separate doses unless the patient experienced disease progression or withdrew consent. Participants had to wait 3 weeks from the last dose of ipilimumab in a parent study to the first dose of ipilimumab in the current study.
  Interventions: Drug: Ipilimumab
- Extended maintenance: Ipilimumab, 0.3 mg/kg (Experimental): Participants who received ipilimumab, 0.3 mg/kg, in a parent study and who achieved extended clinical benefit received the same dose of ipilimumab (0.3 mg/kg) as maintenance in the current study. Maintenance dosing was administered every 12 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipilimumab
- Extended maintenance: Ipilimumab, 3 mg/kg (Experimental): Participants who received ipilimumab, 3 mg/kg, in a parent study and who achieved extended clinical benefit received the same dose of ipilimumab (3 mg/kg) as maintenance in the current study. Maintenance dosing was administered every 12 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipilimumab
- Extended maintenance: Ipilimumab, 10 mg (Experimental): Participants who received ipilimumab, 10 mg/kg, in a parent study and who achieved extended clinical benefit received the same dose of ipilimumab (10 mg/kg) as maintenance in the current study. Maintenance dosing was administered every 12 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipilimumab
- Follow-up (No Intervention): Participants did not receive any additional study treatment in current study but continued follow-up for the collection of survival data.

INTERVENTIONS:
Drug: Ipilimumab — Intravenous solution, 0.3, 3, or 10 mg/kg; 1 dose every 3 weeks or every 3 months until patient discontinuation
  Other Names: BMS-734016; MDX-010
  Arms: Extended maintenance: Ipilimumab, 0.3 mg/kg; Extended maintenance: Ipilimumab, 10 mg; Extended maintenance: Ipilimumab, 3 mg/kg; First reinduction: Ipilimumab, 0.3 to 10 mg/kg; First reinduction: Ipilimumab, 10 to 10 mg/kg; First reinduction: Ipilimumab, 3 to 10 mg/kg

SUMMARY:
The purpose of this study was to evaluate the continued use of ipilimumab in patients who had reinduction at the time of disease progression or to continue maintenance treatment. In addition, this study will continue to follow patients who have taken ipilimumab, but who are not eligible for maintenance or reinduction therapy.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Key Inclusion Criteria

* Diagnosis of advanced melanoma
* Prior treatment in a prespecified prior/parent ipilimumab study
* Men and women 18 years of age and older

First Reinduction:

* No unacceptable toxicity (except select reversible immune-related adverse events) requiring ipilimumab discontinuation
* Had experienced documented progressive disease after expanded clinical benefit

Extended Maintenance

* Received ipilimumab at any dose in a parent study
* Achieved expanded clinical benefit at the time of entry to current study

Follow-up:

* Received ipilimumab at any dose in a closing parent study
* Deemed ineligible for reinduction or extended maintenance treatment or refused treatment as reinduction or extended maintenance at the time of screening in the current study, but consented to follow-up

Key Exclusion Criteria

* Prior treatment with a CD137 agonist or a cytotoxic T-lymphocyte antigen 4 inhibitor or agonist, other than ipilimumab
* Primary ocular or mucosal melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2006-05; Primary Completion 2012-09 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (55):
- United States (19):
  - University Of Arizona Cancer Center, Tucson, Arizona
  - Wilshire Oncology Medical Group Inc, Laverne, California
  - The Angeles Clinic & Research Inst., Los Angeles, California
  - Usc/Norris Comprehensive Cancer Center, Los Angeles, California
  - San Francisco Oncology Associates, San Francisco, California
  - Local Institution, To Come, Connecticut
  - Baptist Cancer Institute, Jacksonville, Florida
  - University Of Chicago, Chicago, Illinois
  - Indiana Oncology Hematology Consultants, Indianapolis, Indiana
  - St Joseph Oncology Inc, Saint Joseph, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Christ Hospital Cancer Center Research, Cincinnati, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Cancer Centers Of The Carolinas, Greenville, South Carolina
  - Center For Oncology Research & Treatment, P.A., Dallas, Texas
  - Joe Arrington Cancer Research And Treatment Center, Lubbock, Texas
  - University Of Washington Medical Center, Seattle, Washington
- Local Institution, Buenos Aires, Buenos Aires, Argentina
- Austria (2):
  - Local Institution, Vienna
  - Local Institution, Wels
- Local Institution, Brussels, Belgium
- Brazil (2):
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Jaú, São Paulo
- Canada (3):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Moncton, New Brunswick
- Local Institution, Olomouc, Czechia
- Local Institution, Aarhus C, Denmark
- France (4):
  - Local Institution, Brest
  - Local Institution, Lyon
  - Local Institution, Paris
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (3):
  - Local Institution, Berlin
  - Local Institution, Heidelberg
  - Local Institution, Kiel
- Israel (2):
  - Local Institution, Jerusalem
  - Local Institution, Tel Aviv
- Italy (4):
  - Local Institution, Genova
  - Local Institution, Meldola (Fc)
  - Local Institution, Rimini
  - Local Institution, Siena
- Local Institution, Oslo, Norway
- Poland (3):
  - Local Institution, Lodz
  - Local Institution, Poznan
  - Local Institution, Wroclaw
- Russia (3):
  - Local Institution, Saint Petersburg
  - Local Institution, Stavropol
  - Local Institution, Voronezh
- South Africa (2):
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Cape Town, Western Cape
- Spain (2):
  - Local Institution, Málaga
  - Local Institution, Valencia
- Local Institution, Dnipro, Ukraine

REFERENCES:
- [Derived] Lebbe C, Weber JS, Maio M, Neyns B, Harmankaya K, Hamid O, O'Day SJ, Konto C, Cykowski L, McHenry MB, Wolchok JD. Survival follow-up and ipilimumab retreatment of patients with advanced melanoma who received ipilimumab in prior phase II studies. Ann Oncol. 2014 Nov;25(11):2277-2284. doi: 10.1093/annonc/mdu441. Epub 2014 Sep 10. PMID 25210016
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 248 enrolled, 6 failed screening; 28 from study CA184-004 (NCT00261365), 42 from CA184-007 (NCT00135408), 67 from CA184-008 (NCT00289627), and 103 from CA184-022 (NCT00289640) entered CA184-025 (NCT00162123). Of enrollees, 2 from study MDX010-08 (NCT00050102) and 6 from MDX010-15 (NCT00729950) entered maintenance as Tumor Assessment Only.
Groups:
- First Reinduction: Ipilimumab, Other Dosage: Participants who received a dose other than 10, 3, or 0.3 mg/kg ipilimumab in parent study received a first reinduction of either 3 or 10 mg/kg in current study.
- Extended Maintenance Only: Ipilimumab, 10 mg/kg: Participants who received ipilimumab, 10 mg/kg, in a parent study and who achieved extended clinical benefit received the same dose of ipilimumab (10 mg/kg) as maintenance in the current study. Maintenance dosing was administered every 12 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
- Extended Maintenance Only: Ipilimumab, 3 mg/kg: Participants who received ipilimumab, 3 mg/kg, in a parent study and who achieved extended clinical benefit received the same dose of ipilimumab (3 mg/kg) as maintenance in the current study. Maintenance dosing was administered every 12 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
- Extended Maintenance Only: Ipilimumab, 0.3 mg/kg: Participants who received ipilimumab, 0.3 mg/kg, in a parent study and who achieved extended clinical benefit received the same dose of ipilimumab (0.3 mg/kg) as maintenance in the current study. Maintenance dosing was administered every 12 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | First Reinduction: Ipilimumab, 10 to 10 mg/kg | First Reinduction: Ipilimumab, 3 to 10 mg/kg | First Reinduction: Ipilimumab, 0.3 to 10 mg/kg | First Reinduction: Ipilimumab, Other Dosage | Extended Maintenance Only: Ipilimumab, 10 mg/kg | Extended Maintenance Only: Ipilimumab, 3 mg/kg | Extended Maintenance Only: Ipilimumab, 0.3 mg/kg | Follow-up
Started | 53 (Enrolled) | 34 (Enrolled) | 24 (Enrolled) | 11 (Enrolled) | 45 (Enrolled) | 13 (Enrolled) | 4 (Enrolled) | 58 (Enrolled)
Received Treatment | 53 | 34 | 24 | 11 | 33 | 12 | 4 | 0
Completed | 9 (Still on treatment) | 5 (Still on treatment) | 3 (Still on treatment) | 3 (Still on treatment) | 14 (Still on treatment) | 4 (Still on treatment) | 0 (Still on treatment) | 0 (Still on treatment)
Not Completed | 44 | 29 | 21 | 8 | 31 | 9 | 4 | 58
Not completed — Disease progression | 27 | 19 | 10 | 4 | 8 | 3 | 1 | 0
Not completed — Study drug toxicity | 6 | 1 | 5 | 0 | 4 | 1 | 1 | 0
Not completed — Death | 3 | 3 | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 1 | 1 | 2 | 1 | 0
Not completed — Deterioration without progression | 2 | 2 | 3 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Not specified (before treatment) | 2 | 0 | 0 | 0 | 12 | 1 | 0 | 0
Not completed — Not specified (after start of treatment) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Tumor assessment only (not treated) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Follow-up only (not treated or assessed) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 57

BASELINE CHARACTERISTICS:
Population: All patients who were enrolled and passed screening in the current study
Groups:
- Extended Maintenance: Ipilimumab, 10 mg/kg: Participants who received ipilimumab, 10 mg/kg, in a parent study and who achieved extended clinical benefit received the same dose of ipilimumab (10 mg/kg) as maintenance in the current study. Maintenance dosing was administered every 12 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | First Reinduction: Ipilimumab, 10 to 10 mg/kg | First Reinduction: Ipilimumab, 3 to 10 mg/kg | First Reinduction: Ipilimumab, 0.3 to 10 mg/kg | First Reinduction: Ipilimumab, Other Dosage | Extended Maintenance: Ipilimumab, 10 mg/kg | Extended Maintenance: Ipilimumab, 3 mg/kg | Extended Maintenance: Ipilimumab, 0.3 mg/kg | Follow-up | Total
Number analyzed (Participants) | 53 | 34 | 24 | 11 | 45 | 13 | 4 | 58 | 242
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.4 (11.7) | 58.8 (9.9) | 56.0 (15.3) | 57.8 (13.7) | 60.5 (12.42) | 59.0 (16.65) | 65.5 (4.80) | 56.3 (12.96) | 57.7 (12.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 11 | 4 | 1 | 20 | 5 | 1 | 22 | 85
  Male | 32 | 23 | 20 | 10 | 25 | 8 | 3 | 36 | 157
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 51 | 34 | 24 | 10 | 45 | 13 | 4 | 55 | 236
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  American Indian/Alaska native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Other: Brazilian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Units on a scale] — ECOG performance status assesses a patient's physical ability against a 6-point scale: 0=fully active, able to carry on all predisease activities without restriction; 1=restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=ambulatory (>50% of waking hours), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead. Score ranges from 0=best status to 5=worst status.
  Units on a scale
    0 | 37 | 22 | 10 | 9 | 40 | 12 | 3 | 29 | 162
    1 | 16 | 11 | 13 | 2 | 5 | 1 | 1 | 10 | 59
    2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3
    3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Not reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With On-study Adverse Events (AEs), AEs Leading to Discontinuation, Serious Adverse Events (SAEs), Drug-related AEs, Immune-related AEs (irAEs), and Death as Outcome
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. An SAE is a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Drug-related is defined as having certain, probable, possible, or missing relationship to study drug. An IrAE is an AE characterized by a potential association with inflammation and considered by the investigator to be drug related. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death.
Time Frame: Continuously from first dose to 70 days after last dose of study drug. For deaths, Day 1 of enrollment to 70 days after last dose of study drug.
Population: All participants who received study drug as reinduction from 0.3, 3, or 10 mg/kg doses in parent study and 10 mg/kg in current study
Measure: Number; unit: Participants
Arm/Group | First Reinduction: Ipilimumab, 10 to 10 mg/kg | First Reinduction: Ipilimumab, 3 to 10 mg/kg | First Reinduction: Ipilimumab, 0.3 to 10 mg/kg
Number analyzed (Participants) | 53 | 34 | 24
Participants
  AEs: Any Grade | 51 | 33 | 24
  AEs: Grade 3 or 4 | 18 | 10 | 10
  AEs: Grade 5 (Fatal) | 4 | 7 | 8
  AEs leading to discontinuation: Any grade | 13 | 6 | 8
  AEs leading to discontinuation: Grade 3 or 4 | 9 | 3 | 6
  AEs leading to discontinuation: Grade 5 (Fatal) | 1 | 2 | 1
  SAEs: Any grade | 23 | 19 | 14
  SAEs: Grade 3 or 4 | 13 | 8 | 5
  SAEs: Grade 5 (Fatal) | 4 | 7 | 8
  Drug-related AEs: Any grade | 42 | 28 | 21
  Drug-related AEs: Grade 3 or 4 | 9 | 3 | 9
  Drug-related AEs: Grade 5 (Fatal) | 0 | 0 | 0
  irAEs: Any grade | 30 | 23 | 18
  irAEs: Grade 3 or 4 | 7 | 2 | 6
  irAEs: Grade 5 (Fatal) | 0 | 0 | 0
  Deaths | 36 | 27 | 19

2. Secondary Outcome: Overall Survival (OS)
Description: OS was computed for all patients who entered this study and is defined as the time between the first dose of study therapy and death. If a patient has not died, OS was censored at the time of last contact.
Time Frame: From first dose of study drug in parent study to death or date of last censoring.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | First Reinduction: Ipilimumab, 10 to 10 mg/kg | First Reinduction: Ipilimumab, 3 to 10 mg/kg | First Reinduction: Ipilimumab, 0.3 to 10 mg/kg
Number analyzed (Participants) | 53 | 34 | 24
Months | 30.8 [24.2 to 41.1] | 18.7 [9.7 to 30.4] | 15.2 [10.7 to 21.4]

3. Secondary Outcome: Percentage of Participants Surviving at 1, 1.5, and 2 Years
Description: Survival rate was defined as the time from first dose of study drug to 1, 1.5, and 2 years.
Time Frame: From first dose of study drug in parent study to up to 2 years after reinduction
Population: All participants who received study drug as reinduction or extended maintenance from 0.3, 3, or 10 mg/kg doses in parent study and 10 mg/kg in current study and those patients who were followed-up.
Measure: Number; unit: Percentage of participants
Groups:
- First Reinduction: Ipilimumab, 0.3 to 10 mg/kg: Participants who initially received ipilimumab, 10 mg/kg, in a parent study received ipilimumab, 0.3 mg/kg in the current study. Ipilimumab was administered as an individual open-label dose every 3 weeks for the first 10 weeks of reinduction for a total of 4 separate doses unless the patient experienced disease progression or withdrew consent. Participants had to wait 3 weeks from the last dose of ipilimumab in a parent study to the first dose of ipilimumab in the current study.
Arm/Group | First Reinduction: Ipilimumab, 10 to 10 mg/kg | First Reinduction: Ipilimumab, 3 to 10 mg/kg | First Reinduction: Ipilimumab, 0.3 to 10 mg/kg | Extended Maintenance: Ipilimumab, 10 mg/kg | Extended Maintenance: Ipilimumab, 3 mg/kg | Extended Maintenance: Ipilimumab, 0.3 mg/kg | Follow-up
Number analyzed (Participants) | 53 | 34 | 24 | 33 | 12 | 4 | 58
Percentage of participants
  1 year | 80.9 | 55.9 | 65.6 | 100 | 100 | 75.0 | 87.8
  1.5 years | 71.3 | 50.0 | 35.0 | 100 | 84.6 | 75.0 | 79.0
  2 years | 63.6 | 38.2 | 30.6 | 91.0 | 84.6 | 75.0 | 64.9

4. Secondary Outcome: Number of Participants With On-study Immune-related Adverse Events (irAEs)
Description: irAEs were defined as adverse events characterized by a potential association with inflammation and considered by the investigator as drug related. These prespecified terms were grouped into the following organ-specific subcategories: gastrointestinal, hepatic, skin, endocrine, neurologic, and other (includes blood, eye, immune system, investigations, infections, renal, and respiratory systems). Patients may have 1 or more events.
Time Frame: From first dose of study drug during reinduction to the earliest of 70 days after last dose or day before second reinduction first dose date
Population: All participants who received study drug as reinduction from 0.3, 3, or 10 mg/kg doses in parent study 10 mg/kg current study
Measure: Number; unit: Participants
Groups:
- First Reinduction: Ipilimumab, 3 to 10 mg/kg: Participants who initially received ipilimumab, 10 mg/kg, in a parent study received ipilimumab, 3 mg/kg in the current study. Ipilimumab was administered as an individual open-label dose every 3 weeks for the first 10 weeks of reinduction for a total of 4 separate doses unless the patient experienced disease progression or withdrew consent. Participants had to wait 3 weeks from the last dose of ipilimumab in a parent study to the first dose of ipilimumab in the current study.
Arm/Group | First Reinduction: Ipilimumab, 10 to 10 mg/kg | First Reinduction: Ipilimumab, 3 to 10 mg/kg | First Reinduction: Ipilimumab, 0.3 to 10 mg/kg
Number analyzed (Participants) | 53 | 34 | 24
Participants
  Any irAE: Any grade | 30 | 23 | 18
  Any irAE: Grade 3 or 4 | 7 | 2 | 6
  Any irAE: Grade 5 (Fatal) | 0 | 0 | 0
  Gastrointestinal irAE: Any grade | 11 | 7 | 14
  Gastrointestinal irAE: Grade 3 or 4 | 2 | 1 | 3
  Hepatic irAE: Any grade | 3 | 0 | 1
  Hepatic irAE: Grade 3 or 4 | 2 | 0 | 1
  Endocrine irAE: Any grade | 3 | 2 | 1
  Endocrine irAE: Grade 3 or 4 | 1 | 0 | 1
  Skin irAE: Any grade | 18 | 18 | 10
  Skin irAE: Grade 3 or 4 | 2 | 1 | 1
  Neurologic irAE: Any grade | 1 | 0 | 0
  Neurologic irAE: Grade 3 or 4 | 0 | 0 | 0
  Other irAE: Any grade | 2 | 3 | 1
  Other irAE: Grade 3 or 4 | 0 | 0 | 0

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time between the date of the baseline tumor assessment in this study and the date of progression or death, whichever occurred first.
Time Frame: From day of first reinduction in current study to date of progression or death, whichever occurred first.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | First Reinduction: Ipilimumab, 10 to 10 mg/kg | First Reinduction: Ipilimumab, 3 to 10 mg/kg | First Reinduction: Ipilimumab, 0.3 to 10 mg/kg
Number analyzed (Participants) | 53 | 34 | 24
Months | 3.4 [2.6 to 7.8] | 2.6 [2.6 to 2.8] | 2.6 [2.0 to 11.1]

ADVERSE EVENTS:
Time Frame: From date of first re-induction first dose to the earliest of 70 days after first re-induction/maintenance last dose date or day before second re-induction first dose date, up to April 2014 (approximately 7 years)
Description: Study initiated: May 2006; Study Completion: April 2014
Arm/Group | First Reinduction: Ipilimumab, 10 to 10 mg/kg | First Reinduction: Ipilimumab, 3 to 10 mg/kg | First Reinduction: Ipilimumab, 0.3 to 10 mg/kg | First Reinduction: Ipilimumab, Other Dosage | Extended Maintenance Only: Ipilimumab, 10 mg/kg | Extended Maintenance Only: Ipilimumab, 3 mg/kg | Extended Maintenance Only: Ipilimumab, 0.3 mg/kg | Follow-up
Serious Adverse Events (participants affected / at risk) | 23/53 | 19/34 | 14/24 | 7/11 | 12/33 | 3/12 | 2/4 | 20/58
Other Adverse Events (participants affected / at risk) | 46/53 | 32/34 | 21/24 | 9/11 | 28/33 | 11/12 | 3/4 | 34/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | First Reinduction: Ipilimumab, 10 to 10 mg/kg (N=53) | First Reinduction: Ipilimumab, 3 to 10 mg/kg (N=34) | First Reinduction: Ipilimumab, 0.3 to 10 mg/kg (N=24) | First Reinduction: Ipilimumab, Other Dosage (N=11) | Extended Maintenance Only: Ipilimumab, 10 mg/kg (N=33) | Extended Maintenance Only: Ipilimumab, 3 mg/kg (N=12) | Extended Maintenance Only: Ipilimumab, 0.3 mg/kg (N=4) | Follow-up (N=58)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 2
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Central nervous system haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 3 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 4 | 0 | 0 | 0 | 0 | 0
Diplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 4 | 5 | 6 | 0 | 0 | 0 | 0 | 12
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endocrine disorder (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient global amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | First Reinduction: Ipilimumab, 10 to 10 mg/kg (N=53) | First Reinduction: Ipilimumab, 3 to 10 mg/kg (N=34) | First Reinduction: Ipilimumab, 0.3 to 10 mg/kg (N=24) | First Reinduction: Ipilimumab, Other Dosage (N=11) | Extended Maintenance Only: Ipilimumab, 10 mg/kg (N=33) | Extended Maintenance Only: Ipilimumab, 3 mg/kg (N=12) | Extended Maintenance Only: Ipilimumab, 0.3 mg/kg (N=4) | Follow-up (N=58)
Abdominal pain (Gastrointestinal disorders) | 7 | 4 | 1 | 0 | 4 | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2 | 0 | 1 | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0 | 1 | 4 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1 | 2 | 1 | 0 | 2
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 5 | 2 | 2 | 0 | 4 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 3 | 0 | 1 | 1 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1 | 1 | 5 | 0 | 0 | 1
Asthenia (General disorders) | 7 | 4 | 1 | 2 | 2 | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 1 | 2 | 4 | 1 | 1 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2
Blood thyroid stimulating hormone increased (Investigations) | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Chills (General disorders) | 6 | 2 | 1 | 0 | 4 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 3 | 0 | 3 | 0 | 4 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 6 | 5 | 4 | 2 | 2 | 1 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 3 | 3 | 7 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 9 | 5 | 5 | 5 | 2 | 2 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 3 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 17 | 8 | 9 | 4 | 16 | 4 | 0 | 3
Dizziness (Nervous system disorders) | 3 | 1 | 1 | 2 | 2 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 3 | 2 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 3 | 1 | 2 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 1
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 20 | 11 | 10 | 6 | 8 | 4 | 1 | 12
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 3 | 2 | 0 | 1 | 0 | 0 | 2
Headache (Nervous system disorders) | 6 | 7 | 1 | 3 | 5 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 4 | 1 | 0 | 0 | 3 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 3 | 1 | 5 | 0 | 0 | 2
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0/1 | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 0 | 3 | 0 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 2 | 1 | 4 | 1 | 0 | 3
Nausea (Gastrointestinal disorders) | 15 | 4 | 7 | 4 | 5 | 2 | 0 | 5
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 3 | 1 | 0 | 0 | 2 | 1 | 0 | 2
Pain (General disorders) | 2 | 0 | 3 | 1 | 2 | 1 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 1 | 2 | 2 | 1 | 6
Photophobia (Eye disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 12 | 6 | 3 | 10 | 3 | 0 | 8
Pyrexia (General disorders) | 5 | 7 | 4 | 0 | 2 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 10 | 10 | 4 | 4 | 6 | 4 | 0 | 6
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 0 | 0 | 5 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 3 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 9 | 2 | 2 | 2 | 2 | 0 | 0 | 1
Weight decreased (Investigations) | 5 | 3 | 4 | 1 | 0 | 0 | 0 | 2
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Significant heterogeneity existed between patients, who rolled over from 6 studies assessing ipilimumab in different doses and combinations. Since not all eligible patients from parent studies were enrolled, some selection bias existed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.